CLINICAL TRIAL: NCT00693979
Title: A Prospective Evaluation in a Randomized Trial of the Safety and Efficacy of the Use of the TAXUS® ElementTM Paclitaxel-Eluting Coronary Stent System for the Treatment of De Novo Coronary Artery Lesions
Brief Title: A Prospective Evaluation in a Randomized Trial of TAXUS in the Treatment of De Novo Coronary Artey Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Boston Scientific Corporation (Industry)
Other Study IDs: Taxus Perseus
Record Dates: First submitted 2008-05-28; First posted 2008-06-09 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TAXUS Element Stent or TAXUS Express Stent — Paclitaxel was selected as the drug to coat the stent because it is known to prevent the uncontrolled cell growth that contributes to the narrowing of artery, by interfering with the ability of cells to divide and multiply. Because of these properties, it has been used as a drug for the treatment of various types of cancer. Cancer patients are given paclitaxel as a solution into the vein. For this study, paclitaxel will be administered locally to the wall of coronary artery as a coating on the stent. Cancer patients receive a dose of paclitaxel approximately 1100 - 1400 times greater than the dose used in the coating of the stent. It is highly unlikely that levels of paclitaxel in the blood would be measurable or have effects anywhere beyond the heart.
  Other Names: Paclitaxel in Taxol; 4.0 mm TAXUS Element stent

SUMMARY:
This study is to compare the safety and performance of two stents coated with the same drug (the TAXUS Element Paclitaxel-Eluting Coronary Stent System and the TAXUS Express2 Paclitaxel-Eluting Coronary Stent System).

DETAILED DESCRIPTION:
Approximately 1264 subjects at a maximum of 100 clinical sites will be part of this study. This study will recruit approximately 30 subjects from NHC & NUH (12 from NUH) over a period of 6 to 9 months recruitment period.

Paclitaxel is the active ingredient in Taxol®, a drug originally developed to treat cancer. The addition of the paclitaxel coating to the stent could improve the performance of the stent by preventing the re-narrowing of the treated coronary artery. This re-narrowing is called restenosis. Restenosis can occur after balloon angioplasty or the placement of a stent and is the result of too much cell growth at the treatment site in the coronary artery.

The TAXUS Element stent is an investigational device. The term investigational means that the stent is not currently approved for commercial use by the FDA or other regulatory agencies worldwide. The TAXUS Express 2 stent is also a coronary stent made with the same drug coating as the Element stent. It is approved for commercial use by the FDA and other regulatory agencies worldwide, with the exception of the 4.0 mm size, which is not yet approved by the FDA. However, the 4.0 mm size was studied for safety and performance in a clinical trial and the results of that trial have been submitted to FDA to support approval. FDA has agreed that the 4.0 mm size may be used in this trial.

Paclitaxel was selected as the drug to coat the stent because it is known to prevent the uncontrolled cell growth that contributes to the narrowing of artery, by interfering with the ability of cells to divide and multiply. Because of these properties, it has been used as a drug for the treatment of various types of cancer. Cancer patients are given paclitaxel as a solution into the vein. For this study, paclitaxel will be administered locally to the wall of coronary artery as a coating on the stent. Cancer patients receive a dose of paclitaxel approximately 1100 - 1400 times greater than the dose used in the coating of the stent. It is highly unlikely that levels of paclitaxel in the blood would be measurable or have effects anywhere beyond the heart.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria

* Subject is ≥ 18 years old and ≤ 80 years old
* Eligible for percutaneous coronary intervention (PCI)
* Documented stable angina pectoris (Canadian Cardiovascular Society [CCS] Classification 1, 2, 3, or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
* Acceptable candidate for coronary artery bypass grafting (CABG)
* Left ventricular ejection fraction (LVEF) is > 30%
* Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
* Subject willing to comply with all specified follow-up evaluations

Angiographic Inclusion Criteria (visual estimate)

* Target lesion located in native coronary artery
* Target lesion must be de novo
* Target lesion diameter stenosis > 50%
* Reference vessel diameter (RVD) > 2.75mm to < 4.0mm
* Cumulative target lesion length < 28 mm (area to be treated must be completely coverable by one study stent)
* Target lesion is successfully pre-dilated. Subjects are enrolled after successful balloon catheter pre-dilation of the target lesion and assignment to treatment arm by IVRS.
* One non-target lesion may be treated in a non-target vessel
* Non-target lesion in non-target vessel must be treated with a commercially available TAXUS stent if use of drug-eluting stent required.
* Treatment must be deemed a clinical angiographic success, without requiring use of unplanned additional stent(s).
* Treatment must be completed prior to treatment of target lesion.

Exclusion Criteria:

Clinical Exclusion Criteria

* Contraindication to ASA, or to both clopidogrel and ticlopidine
* Known hypersensitivity to paclitaxel
* Known allergy to stainless steel
* Known allergy to platinum
* Previous treatment of the target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent
* Previous treatment of the target vessel with a bare metal stent (BMS) within 9 months of the index procedure
* Previous treatment of any non-target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent within 9 months of the index procedure
* Previous treatment with intravascular brachytherapy in the target vessel
* Planned PCI or CABG post-index procedure
* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement
* Myocardial infarction (MI) within 72 hours prior to the index procedure as defined per protocol definition (see Appendix A)
* Cerebrovascular accident (CVA) within the past 6 months
* Cardiogenic shock characterized by systolic pressure < 80mm Hg and/or central filling pressure > 20 mm Hg, or cardiac index < 1.8 liters/minute/m2 or intra-aortic balloon pump or intravenous inotropes are needed to maintain a systolic pressure > 80 mm Hg and a cardiac index > 1.8 liters/minute/m2
* Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl or 177 μmol/l)
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure
* Leukopenia (leukocyte count < 3.5 x 109/liter)
* Thrombocytopenia (platelet count < 100,000/mm3)
* Thrombocytosis (> 750,000/mm3)
* Active peptic ulcer or active gastrointestinal (GI) bleeding
* Current treatment, or past treatment within 12 months of the index procedure, with paclitaxel or other chemotherapeutic agent(s)
* Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9 months after the index procedure
* Male or female with known intention to procreate within 9 months after the index procedure
* Positive pregnancy test within 7 days before the index procedure, or lactating
* Life expectancy of less than 24 months due to other medical conditions
* Co-morbid condition(s) that could limit the subject's ability to comply with study follow-up requirements or impact the scientific integrity of the study
* Currently participating in another investigational drug or device study

Angiographic Exclusion Criteria (visual estimate)

* Target lesion in left main artery, whether protected or unprotected
* Target lesion is a chronic total occlusion (TIMI flow < 1)
* Target lesion is restenotic
* Target lesion is located in a saphenous vein graft or mammary artery graft
* Target lesion is accessed via saphenous vein graft or mammary artery graft
* Target lesion is < 5mm from bare metal stent (BMS)
* Target lesion is < 5mm from ostium
* Target lesion is < 5 mm from a side branch vessel ≥ 1.5 mm in diameter
* Untreated lesions with ≥ 50% diameter stenosis or thought to impair flow remaining in target vessel
* Target lesion and/or target vessel proximal to the target lesion is moderately or severely calcified
* Target lesion and/or target vessel proximal to the target lesion is severely tortuous
* Target lesion is located within or distal to a > 60° bend in the vessel
* Target lesion with angiographic presence of probable or definite thrombus
* Unprotected left main coronary artery disease
* Protected left main coronary artery disease with target lesion in LAD or LCx(subject may be enrolled if only lesion is target lesion in RCA)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult